CLINICAL TRIAL: NCT02911077
Title: Longitudinal Changes in the Oral and Gut Microbiome of Individuals With Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160162; 16-CC-0162
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Alcoholic Intoxication; Alcohol-Related Disorders
Keywords: Bacteria; Natural History
MeSH Terms: conditions — Alcoholic Intoxication; Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AUD population: The participants/group were treatment-seeking AUD individuals admitted to the NIH CC 1SE Addictions Unit.

SUMMARY:
Background:

Many bacteria live in the gut. The gut is the tube that moves food from the mouth through the stomach to the intestines. Heavy alcohol use disturbs these bacteria. There is evidence that the bacteria in the gut may affect anxiety and depression. Researchers want to learn more about these bacteria in order to better treat diseases such as alcohol dependence.

Objective:

To identify the different bacteria that live in the mouth and gut. Also, to learn if these bacteria change as a person goes through alcohol detoxification.

Eligibility:

People ages 18 and older who:

* Enrolled in screening protocol 14-AA-0181
* Are going through detoxification treatment at the Clinical Center

Design:

Participants will have physical exams.

Participants will answer questions about:

* Anxiety and depression
* Alcohol use
* Sleep
* Abdominal and oral health
* Diet

Participants will keep a regular record of their diet.

Participants will have breath alcohol analysis 4 times per day.

Participants will provide stool and oral specimens at most once a day for the first week. Then, they will provide them once a week while they are at the Clinical Center.

* For the oral specimen: A small brush rubs the tongue. They may not eat, drink, or perform oral care within 2 hours of collection.
* For the stool specimen: They will receive a container that fits in the toilet. They will let the nurse know right away when the sample is ready.

Participants will have a dental visit. This consists of an oral exam and oral health assessment. The dentist may recommend a cleaning or dental X-rays.

DETAILED DESCRIPTION:
The microbiome exists in a complex symbiotic relationship with its human host, the characterization of which is imperative for understanding a myriad of diseases. Until recently, much of gut microbiome research has focused on gastrointestinal disorders. Recent research, however, has implicated the gut microbiome in psychological disorders as well through a proposed gut-brain axis. Of particular interest is characterization of the microbiome of individuals with severe alcohol use disorders, as alcohol has been known to profoundly alter the gut microbiome. For many years, scientists have theorized a connection between the proinflammatory mediators produced by ethanol consumption, liver disease and the gut microbiome. This study represents the first instance in which the naturalistic time course of changes in the gut microbiome will be followed in alcoholics in whom detailed history of alcohol consumption and diet have been obtained. We hypothesize that the gut microbiome will renormalize spontaneously and without specific intervention over a time frame of one or two weeks. Alcoholic patients also suffer from serious oral hygiene problems associated with alterations in oral microbial flora. We hypothesize that abnormalities in the oral microbiome will be detectable on admission, and that these will also rapidly renormalize with abstinence and resumption of ordinary diet and oral hygiene. If not, the findings in this study could point to the need for other interventions, such as administration of probiotics. Twenty evaluable participants admitted to the Clinical Center for alcohol detoxification will be enrolled. All patients will be admitted under the Unit and Clinic Evaluation, Screening, Assessment, and Management protocol (14-AA-0181), which includes adults 18 years of age or older seeking treatment for severe alcohol use disorders. Oral (tongue brushings) and gut (stool) specimens will be collected daily for the first week and then once a week for 28 days. Demographic characteristics, detailed drinking and dietary histories, measures of addiction severity, comorbid mental disorders, and metabolic indicators of other disease will be collected for correlation with microbiological results. Dietary records will include use of probiotics. Exclusion criteria include use of antibiotics, corticosteroids or immunosuppressive agents within the past month. Informed consent will be obtained after consent for the screening and treatment protocol (14-AA-0181) and in accordance with policies protecting participants with impaired decision-making. Microbial identification will include 16S rRNA analysis and a validated Next Generation Sequencing analysis pipelines. Statistical comparisons between each patient's oral and gut microbiome samples will be evaluated and all results from this population will also be compared to published microbiomes in both healthy volunteers as well as existing data from alcohol dependent individuals. Participants will be compensated for research-related discomfort and inconveniences in accordance with NIH guidelines.

ELIGIBILITY:
* INCLUSION CRITERIA:
* At least 18 years of age
* Willing to provide consent
* Consented on screening and research protocol 14-AA-0181
* Admitted to the NIH CC for inpatient detoxification treatment

EXCLUSION CRITERIA:

* Currently using or have used any of the following drugs within the last month by self-report:

  * Antibiotics
  * Corticosteroids: inhaled, oral, intravenous or intramuscular
  * Immunosuppressive or cytotoxic agents
* Large doses of probiotics such as supplemental probiotics (ordinary dietary components such as beverages/milk or yogurt DO NOT APPLY)
* Major surgery of the GI tract with the exclusion of cholecystectomy and appendectomy in the past 5 years.
* Any bowel resection at any time.
* History of active uncontrolled gastrointestinal disorders or diseases including inflammatory bowel disease, ulcerative colitis, Crohn s disease, and/or infectious gastroenteritis, colitis, or gastritis (per patient s report of whether or not they have been diagnosed by a physician).
* Enrolled in any investigational study that might affect the microbiome.
* BMI greater than or equal to 30 kg/m2

Some of these exclusionary criteria have been adapted from the Human Microbiome Project [40]. All exclusion measures will be collected from self-report.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatient treatment seeking alcohol dependent participants
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Identification of bacteria in the gut and oral microbiomes over time | all timepoints
  Characterization of the gut and oral micro biome

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Maki, C.R.N.P., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0162.html